CLINICAL TRIAL: NCT02796235
Title: Prospective and Monocentric Study of the Incidence of Venous Thromboembolic Disease (VTE) in Spinal Cord Injury (SCI) Patient Between 3 and 12 Months After SCI
Acronym: IMATEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC12_0137
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal cord injury (SCI) patient (Other)
  Interventions: Other: Venous Doppler ultrasound of the lower limbs

INTERVENTIONS:
Other: Venous Doppler ultrasound of the lower limbs — Venous Doppler ultrasound of the lower limbs at 6, 9 and 12 months of the initial injury

SUMMARY:
Venous Thromboembolic Disease (VTE) in SCI patients is very common, its prevalence is 60 to 80% against 10-20% in the general population.

The risk of VTE is very important in the first weeks after spinal cord injury, and then declines with a prevalence of VTE slightly higher than the general population after 12 weeks. However there is no prospective study of incidence of VTE in SCI patients after 3 months. The investigators wish to conduct such a study during the year following spinal cord injury with performing venous Doppler ultrasound of the lower limbs 6, 9 and 12 months of the initial injuryassociated with a standardized clinical assessment, to know the incidence of VTE and determine prognostic factors for VTE.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Patients having paraplegia or tetraplegia from C2 levels and above S1
* Paraplegia and tetraplegia of traumatic or non progressive SCI from traumatic or medical origin (ischemic, post-surgical, myelitis, benign tumor)
* Informed consent signed.
* stabilized respiratory situation with absence of chronic hypoxemia (hypoxemia being characterized by PaO2 steady state <7.33 kPa)
* Patient not amputated.
* Absence of heart failure with ejection fraction below 30%
* Lack of solid neoplasia or progressive lymphoid haemopathy for 5 years, or myeloproliferative disorders (including polycythemia and thrombocythemia).
* No personal history of VTE and / or thrombophilia before the injury.

Exclusion Criteria:

* Unstabilized respiratory situation with presence of chronic hypoxemia (hypoxemia being characterized by PaO2 steady state <7.33 kPa)
* Amputated Patient.
* Patients with heart failure with ejection fraction below 30%
* Solid neoplasia or progressive lymphoid haemopathy for 5 years, or myeloproliferative disorders (including polycythemia and thrombocythemia).
* Personal history of VTE and / or thrombophilia before the injury.
* Can not to follow during the study period
* Pregnant women
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Number of appearances of phlebitis in the lower limbs and / or pulmonary embolism in spinal cord injury (SCI) patient between 3 and 12 months after SCI | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No